CLINICAL TRIAL: NCT03962114
Title: Effects of Nicotinamide Riboside (Vitamin B3) in Patients With Ataxia Telangiectasia.
Brief Title: Effects of Vitamin B3 in Patients With Ataxia Telangiectasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: A-T Children's Project (Other); Twan foundation (https://twanfoundation.nl) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL68197.091.18
Record Dates: First submitted 2019-04-11; First posted 2019-05-23 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2019-03

CONDITIONS: Ataxia Telangiectasia; ATM Gene Mutation
Keywords: Ataxia Telangiectasia; ATM Gene Mutation; ATM protein; Nicotinamide riboside
MeSH Terms: conditions — Ataxia Telangiectasia; Hereditary Sensory and Autonomic Neuropathies | interventions — Niacinamide; nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Open label proof of concept study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention group (Experimental): treatment with vitamin B3
  Interventions: Dietary Supplement: Vitamin B3

INTERVENTIONS:
Dietary Supplement: Vitamin B3 — capsules with niagen
  Other Names: Nicotinamide riboside

SUMMARY:
This clinical trial investigates the effects of nicotinamide riboside (vitamin B3) on the disease course of patients with ataxia telangiectasia.

Patients will be treated during four consecutive months with nicotinamide riboside (25mg/kg/day), followed by a washout period of two months.

Main study parameters/endpoints: Ataxia, dysarthria, quality of life, laboratory parameters.

DETAILED DESCRIPTION:
Rationale: Ataxia Telangiectasia (A-T) is an autosomal recessively inherited neurodegenerative disorder, with a high cancer risk, that also affects the immune and respiratory system. Therapy for A-T is restricted to symptomatic treatment including rehabilitation care, combined with infection prevention and treatment, and screening for pulmonary dysfunction and malignancies. A-T is caused by mutations in the ATM gene. The ATM protein plays a pivotal role in more than 100 different biochemical processes, among which cellular energy metabolism, cell signaling, and DNA repair. Nicotinamide adenine dinucleotide (NAD+) is an essential molecule in many of these processes and studies have shown that NAD+ deficiency plays a role in disease mechanisms underlying DNA repair disorders such as A-T. NAD+ is available in food, but can also be synthesized in the body from its precursors nicotinamide, nicotinic acid, and nicotinamide riboside (NR), as a group called "vitamin B3". Treatment of experimental A-T animal models with NR showed beneficial effects. The aim of this study is to investigate whether treatment with NR during a period of six months may have positive effects on the disease course of patients with A-T.

Objective: To investigate the effects of NR on the disease course of patients with ataxia telangiectasia.

Study design: Single center, interventional, explorative, open-label proof of concept study.

Study population: Patients with A-T (age >2 years).

Intervention (if applicable): Patients will be treated with nicotinamide riboside (25mg/kg/day), during four consecutive months, followed by a washout period of two months.

Main study parameters/endpoints: Ataxia, dysarthria, quality of life, laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* A-T patients who visit our outpatient clinic.
* Genetically confirmed diagnosis of A-T by the identification of pathogenic mutations of the ATM gene.
* Age ≥ 2 years or older and bodyweight ≥ 12 Kg.
* Informed consent.

Exclusion Criteria:

* Additional medical condition or illness that impair the patient's ability to participate in the study (e.g. actual treatment of a malignancy, active infection, poorly controlled diabetes mellitus, hypertension, organ failure, clinically significant hematological or biochemical abnormalities different from the usual abnormalities in A-T)
* Elevated serum transaminases (> 2 times upper limit of normal)
* Participation in another interventional study at start of the study or during the study
* Pregnancy.
* Breast feeding.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Ataxia, SARA (Scale of the assesment and rating of ataxia) | change from baseline -1 month - 4 months - 6 months
  Changes in the total score will be measured.
Ataxia, ICARS (International Cooperative Ataxia Rating Scale) | change from baseline -1 month - 4 months - 6 months
  Changes in the total score will be measured.
Ataxia, 9-hole pegboard test. | change from baseline -1 month - 4 months - 6 months
  Changes in fastes time of the 9-hole pegboard test will be measured.
Dysarthria, Radboud dysarthria assesment (RDA) | change from baseline -1 month - 4 months - 6 months
  Changes in maximum performance tasks and severity of dysarthria will be measured.

SECONDARY OUTCOMES:
Quality of life questionnaire EuroQoL 5 Dimensions 5 Levels (EQ-5D-5L) | change from baseline -1 month - 4 months - 6 months
  Changes in the total quality of life score will be measured.
Laboratory measurements | change from baseline -1 month - 4 months - 6 months
  Results will be summarized descriptively, with abnormal and clinically notable values/findings being identified
Intelligibility, Intelligibility in Context Scale (ICS) | change from baseline -1 month - 4 months - 6 months
  Changes in the total score of the Intelligibility in Context Scale (ICS), will be measured.
Fatigue, Visual Analogous Scale (VAS) | change from baseline -1 month - 4 months - 6 months
  Changes in the total VAS score will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Willemsen, Prof., Principal Investigator — michel.willemsen@radboudumc.nl
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No